CLINICAL TRIAL: NCT03030053
Title: Mechanistic Assessment of the Acute and Chronic Cognitive Effects of Flavanol/Anthocyanin Intervention in Humans - Chronic Trial
Brief Title: The Effects of Flavonoid Supplementation on Cognition and Neural Mechanisms in Healthy Older Adults
Acronym: CoCo_Chronic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Reading (Other)
Collaborators: Mars, Inc. (Industry); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Nutritional Medicine, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UREC1548_CoCo_ChronicTrial
Record Dates: First submitted 2016-05-07; First posted 2017-01-24 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Mental Processes
Keywords: Flavanols; Flavonoids; Polyphenols; Cognition; Aging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Cocoa-Flavanol Supplements: 3 capsules per day each containing 300mg (total dose of 900mg daily) for 24 weeks
  Interventions: Dietary Supplement: Cocoa-Flavanol Supplements
- Control (Placebo Comparator): Control Supplements: 0mg cocoa-flavanols per day for 24 weeks
  Interventions: Dietary Supplement: Control Supplements

INTERVENTIONS:
Dietary Supplement: Cocoa-Flavanol Supplements — 3 capsules each containing 300mg cocoa flavanols (total daily dose of 900mg cocoa-flavanols).
  Arms: Active
Dietary Supplement: Control Supplements — 3 capsules each containing 0mg cocoa-flavanols
  Arms: Control

SUMMARY:
A double-blind, randomised, controlled, parallel arm chronic intervention trial with healthy older adults will be conducted to determine the effect of a flavonoid-rich supplement on cognitive function, peripheral arterial health and brain mechanisms. It is predicted that chronic flavonoid supplementation will result in cognitive benefits and that these may be due to beneficial effects of flavonoids on vascular and brain function.

DETAILED DESCRIPTION:
There has recently been an increasing interest in the potential of flavonoids, plant derived compounds found in foods such as fruit and vegetables, to improve cognitive function. Research suggests that flavonoids improve memory and learning, possibly as a result of their anti-inflammatory and neuroprotective effects, for example by increasing cerebral blood flow (CBF), protecting vulnerable neurons, or by stimulating neuronal function and growth. The proposed research will involve a parallel design chronic dietary supplementation trial using a flavonoid-supplement and a matched control containing no flavonoids, to investigate long-term changes in cognitive performance. To understand the neural mechanisms behind potential changes in cognitive performance, resting cerebral blood flow (CBF), blood-oxygen level dependent (BOLD) response during two sensitive tests of cognitive performance, and structural brain changes will be measured in a group of healthy elderly adults (N=70, age range 60-75 years) using magnetic resonance imaging (MRI). Additionally, peripheral vascular health will be measured using flow mediated dilatation (FMD), and bioavailability of flavonoid monomers and metabolites will be determined through analysis of plasma and urine samples. Biomarkers in the blood associated with vascular health and neural functioning as well as markers of interest in relation to the possible mechanisms of action of flavonoids will also be measured. All endpoints will be acquired before and after a 24-week chronic supplementation of either a high flavonoid supplementation or a control product, consumed in addition to participants' normal diet. Measures will also be taken following a 12-week post-intervention washout period in order to investigate whether any beneficial effects are sustained following cessation of supplementation.

ELIGIBILITY:
INCLUSION CRITERIA:

* Males and females aged 60-75 years
* English as primary language, able to understand the study information sheet, follow instructions in English and give informed consent
* Non-smokers
* Alcohol consumption should be within the current National Health Service (NHS) recommendation - women: ≤21 units per week (max 3 per day), 1 large 250mL glass of wine (Alcohol By Volume 12%) is 3 units; men: ≤ 28 units per week (max 4 per day), 1 pint of strong lager/beer/cider (Alcohol By Volume 5.2%) is 3 units
* BP <150/90 (determined at screening)
* BMI <30 (determined at screening)
* Full blood count parameters within the normal range, specifically:

  * Haemoglobin to check for anaemia (>12.5 g/dL for males and >11.5 g/dL for females)
  * Total white cell count (3.6-11.0 x109/L)
  * Differential count:

    * Neutrophils (1.8 - 7.5 x109/L)
    * Lymphocytes (1.0 - 4.0 x109/L)
    * Monocytes (0.2 - 0.8 x109/L)
    * Eosinophils (0.1 - 0.4 x109/L)
    * Basophils (0.02 - 0.1 x109/L)
  * Normal platelet function (platelet count 140-400 x109/L)
  * Red cell count (4.50-6.50 x1012/L for males; 3.80-5.80 x1012/L for females)
  * Haematocrit (0.40-0.54 L/L for males; 0.37-0.47 L/L for females)
  * Mean Cell Volume (80-100 fL)
  * Mean Cell Haemoglobin (27-32 pg)
  * Reticulocyte Count (0.2-2.0 %)
* The following blood parameters within the normal range:

  * Liver function (gamma-glutamyl transpeptidase [GGT] level < 80 IU/L, alanine transaminase [ALT] < 30 U/L, alkaline phosphatase [ALP] < 320 U/L),
  * Kidney function (total bilirubin ≤ 22 μmol/L, creatinine ≤ 106 μmol/L, uric acid < 506 μmol/L),
  * Fasting blood glucose level (< 7 mmol/L),
  * Triglycerides (< 2.2 mmol/L)
  * Plasma cholesterol (< 8 mmol/L)

EXCLUSION CRITERIA:

* General global cognitive impairment (Mini Mental State Examination score < 24)
* Un-corrected vision or hearing problems
* Speech or communication difficulties
* Currently suffering from depression (Brief Symptom Inventory score of ≥ 11)
* Diagnosed with any learning difficulty such as Dyslexia or Dyspraxia
* Sensitive/allergic to the intervention or any of the study foods
* Suffering from any form of clinically diagnosed disease, including:

  * Major mental illness (current or previous episode with hospitalization)
  * Chronic fatigue syndrome
  * Liver disease
  * Diabetes mellitus
  * Heart disease or myocardial infarction
* Taking blood pressure medication, anticoagulants, anti-platelet medication or antidepressants
* On a weight reducing dietary regimen or taking any dietary supplements (including dietary fatty acids), unless willing to temporarily refrain from taking dietary supplements for the duration of the study
* Subjects consuming more than seven portions of fruit and vegetables a day
* Subjects consuming more than five cups of tea a day
* Men taking part in more than 10.5 hours of moderate to vigorous exercise per week and women taking part in more than 7 hours of moderate to vigorous exercise per week (assessed on an individual basis to avoid recruitment of people who exercise too vigorously)
* Taking illegal substances

MRI part:

* Has a heart pacemaker or metal implants (including any non-removable ferro-magnetic dental items)
* Any body piercing items that cannot be removed
* Is claustrophobic

Note: Participation in other research trials within the last month will need to be declared and may affect the start date for participation in the current trial.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Performance (0-24 weeks) | Change from baseline (pre intervention) to week 24 (post intervention)
  Composite measure of global cognitive function (scores from different cognitive tasks will be standardised to allow an overall score of global cognitive function to be calculated)
Change in Cognitive Performance (0-36 weeks) | Change from baseline (pre intervention) to week 36 (follow-up)
  Composite measure of global cognitive function (scores from different cognitive tasks will be standardised to allow an overall score of global cognitive function to be calculated)

SECONDARY OUTCOMES:
Change in Flow Mediated Dilatation (0-24 weeks) | Change from baseline (pre intervention) to week 24 (post intervention)
  Technique to measure the flexibility of the endothelium in larger peripheral blood vessels
Change in Flow Mediated Dilatation (0-36 weeks) | Change from baseline (pre intervention) to week 36 (follow-up)
  Technique to measure the flexibility of the endothelium in larger peripheral blood vessels
Change in cerebral blood flow (0-24 weeks) | Change from baseline (pre intervention) to week 24 (post intervention)
  Use of arterial spin labelling to determine cerebral blood flow at rest
Change in cerebral blood flow (0-36 weeks) | Change from baseline (pre intervention) to week 36 (post intervention)
  Use of arterial spin labelling to determine cerebral blood flow at rest
Change in brain activity (0-24 weeks) | Change from baseline (pre intervention) to week 24 (post intervention)
  Use of functional MRI to determine BOLD response (indicative of brain activation) during cognitive activity
Change in brain activity (0-36 weeks) | Change from baseline (pre intervention) to week 36 (post intervention)
  Use of functional MRI to determine BOLD response (indicative of brain activation) during cognitive activity
Change in brain structure (0-24 weeks) | Change from baseline (pre intervention) to week 24 (follow-up)
  Use of high resolution images to determine changes to brain structure such as grey and white matter
Change in brain structure (0-36 weeks) | Change from baseline (pre intervention) to week 36 (follow-up)
  Use of high resolution images to determine changes to brain structure such as white and grey matter
Change in flavanol monomer levels | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of epicatechin and catechin in plasma and urine samples
Change in procyanidin levels | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of procyanidin dimers through to decamers in plasma and urine samples
Change in levels of flavanol monomer metabolites/derivatives | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of epicatechin and catechin metabolites/derivatives in plasma and urine samples
Change in levels of procyanidin metabolites/derivatives | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of procyanidin metabolites/derivatives in plasma and urine samples
Change in levels of nitroso compounds | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of nitric oxide, nitrate and nitrite levels in plasma/serum &/ urine
Change in levels of markers of inflammation | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of pro and anti-inflammatory cytokines and C-reactive protein (CRP) levels in plasma/serum
Change in levels of markers of neuronal function | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of brain-derived neurotrophic factor (BDNF) and lactate in plasma/serum
Change in levels of a marker of stress/anxiety | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of cortisol in plasma/serum
Change in levels of a marker of oxidative stress | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of uric acid in plasma/serum
Change in levels of markers of vascular function/cardiovascular disease (CVD) risk | Change from baseline (pre intervention) to week 24 (post intervention)
  Concentrations of glucose, insulin, cholesterol (total, high density lipoprotein [HDL], low density lipoprotein [LDL]), non-esterified fatty acids [NEFA], triglycerides [TAG] in plasma/serum

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
To achieve the aim of data sharing with the wider community data will be submitted for inclusion in the Biotechnology and Biological Sciences Research Council (BBSRC)-funded Code Analysis, Repository & Modelling for E-Neuroscience (CARMEN) depository for neurophysiological datasets (http://www.carmen.org.uk). Data will also be accessible by making a direct request to the PI, and will be transferred to the recipient. Publications will be in open access journals where possible. If not possible, due to the need to reach the widest possible audience, pre-publication manuscripts arising from the project will be deposited in the free and publicly searchable University of Reading research database (CentAUR: http://centaur.reading.ac.uk). All data will be made available in an anonymised format upon request following publication of main findings. It is envisaged that the entire datasets will be available 6 months following the end of the project and maintained for a period of at least 10 years.